CLINICAL TRIAL: NCT03067948
Title: Improving Identification of Mental Health/Substance Use Disorders in HIV Primary Care: Pilot Clinical Response
Acronym: PROACT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: IRB00115401; 5K23MH105284 (NIH)
Record Dates: First submitted 2016-12-06; First posted 2017-03-01 (Actual); Results first posted 2018-11-19 (Actual); Last update posted 2018-11-19 (Actual); Status verified 2018-11

CONDITIONS: HIV Infections
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention - Positive Screen Shared (Experimental): In the intervention, participants will be given the opportunity to determine which positive screen, if any, that the participant would like to discuss with the participant's provider at the next HIV primary care appointment. The participant will be notified that all positive screens will be shared with the provider prior to the participant's next HIV primary care visit, and that any positive screen the patient has chosen to discuss with the provider will be specified. The provider will receive the PROs result (score, interpretation, and recommendation) prior to the next HIV primary care visit.
  Interventions: Behavioral: Patient Designated Positive Screen Shared with Provider

INTERVENTIONS:
Behavioral: Patient Designated Positive Screen Shared with Provider — Patient Designated Positive Screen Shared with Provider -- In the intervention, participants will be given the opportunity to determine which positive screen, if any, that the participant would like to discuss with the participant's provider at the next HIV primary care appointment. The participant will be notified that all positive screens will be shared with the provider prior to their next HIV primary care visit, and that any positive screen the patient has chosen to discuss with the provider will be specified. The provider will receive the PROs result (score, interpretation, and recommendation) prior to their next HIV primary care visit

SUMMARY:
This research is a feasibility pilot of an intervention to respond to positive screening tests for mental health(MH) and substance use (SU) captured through the Patient Reported Outcomes questionnaires (PROs). The PROs are currently performed in the clinic, however, the results are neither reviewed with patients nor transmitted to providers. This pilot assesses the feasibility of moving the PROs into the clinical realm by having patients review the PRO results, identifying an issue to discuss at the patient's next HIV primary care visit, and determining whether this process increases discussion of MH and SU disorders in the subsequent clinical visit and/or increases referrals to MH and/or SU treatment.

ELIGIBILITY:
Inclusion Criteria:

* must be enrolled in the Johns Hopkins Clinical Cohort at the Johns Hopkins Moore Clinic
* must be living with HIV

Exclusion Criteria:

-

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2017-02-09 (Actual); Primary Completion 2017-06-30 (Actual); Study Completion 2017-07-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anne Monroe, MD, MSPH, Principal Investigator — Johns Hopkins University
Locations (1):
- Moore Clinic for HIV Care, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: We only enrolled an intervention group (and utilized a historic control). Thus, all patient participants were assigned to the intervention group.
Groups:
- Intervention - Positive Screen Shared: Participants were given the opportunity to determine which positive screen, if any, that the participant wanted to discuss with the participant's provider at the next HIV primary care appointment. The participant was notified that all positive screens would be shared with the provider prior to the participant's next HIV primary care visit, and that any positive screen the patient chose to discuss with the provider would be specified. The received the Patient Reported Outcomes (PROs) result (score, interpretation, and recommendation) prior to the next HIV primary care visit.
Period: Overall Study
Arm/Group | Intervention - Positive Screen Shared
Started | 32
Completed | 32
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Intervention - Positive Screen Shared: In the intervention, participants were given the opportunity to determine which positive screen, if any, that the participant would like to discuss with the participant's provider at the next HIV primary care appointment. The participant was notified that all positive screens will be shared with the provider prior to the participant's next HIV primary care visit, and that any positive screen the patient had chosen to discuss with the provider will be specified. The provider received the PROs result (score, interpretation, and recommendation) prior to the next HIV primary care visit.
Arm/Group | Intervention - Positive Screen Shared
Number analyzed (Participants) | 32
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.6 (8.9)
Sex/Gender, Customized [Number; unit: participants]
  Male | 21
  Female | 11
Race/Ethnicity, Customized [Number; unit: participants]
  Black | 29
  White | 2
  Other | 1

OUTCOME MEASURES:

1. Primary Outcome: Mental Health or Substance Use Issue Raised in Visit
Description: Number of participants for whom review and coding of audio recording captured a mental health or substance use issue during their visit
Time Frame: Visit following intervention which will occur on the same day or up to 1 week after the intervention
Measure: Count of Participants; unit: Participants
Groups:
- Intervention - Positive Screen Shared: Participants were given the opportunity to determine which positive screen, if any, that the participant wanted to discuss with the participant's provider at the next HIV primary care appointment. The participant was notified that all positive screens would be shared with the provider prior to the participant's next HIV primary care visit, and that any positive screen the patient chose to discuss with the provider would be specified. The received the PROs result (score, interpretation, and recommendation) prior to the next HIV primary care visit.
Arm/Group | Intervention - Positive Screen Shared
Number analyzed (Participants) | 32
Participants | 32

2. Primary Outcome: Audio Recording Data - Mental Health/Substance Use Action Taken
Description: Number of participants for whom review of transcript of clinic visit characterized discussion of mental health issues and referral for services
Time Frame: Visit following intervention which will occur on the same day or up to 1 week after the intervention
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention - Positive Screen Shared
Number analyzed (Participants) | 32
Participants | 32

ADVERSE EVENTS:
Time Frame: intervention consisted of 1 study visit; no subsequent monitoring of participants was undertaken
Description: The intervention only lasted the duration of the study visit; no subsequent monitoring was performed.
Arm/Group | Intervention - Positive Screen Shared
All-Cause Mortality (participants affected / at risk) | 0/32
Serious Adverse Events (participants affected / at risk) | 0/32
Other Adverse Events (participants affected / at risk) | 0/32

LIMITATIONS AND CAVEATS:
The sample size was small and recruited patients from one urban outpatient infectious diseases clinic, and may not be generalizable to other patient populations living with HIV.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-12-20): https://cdn.clinicaltrials.gov/large-docs/48/NCT03067948/Prot_SAP_000.pdf